CLINICAL TRIAL: NCT00663858
Title: Cetrorelix Pamoate (AEZS-102) in Patients With Symptomatic BPH: a Double-blind Placebo-controlled Efficacy Study
Brief Title: Cetrorelix Pamoate in Patients With Symptomatic Benign Prostatic Hypertrophy (BPH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEZS-102-036
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Results first posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2010-12

CONDITIONS: Benign Prostatic Hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cetrorelix 78+78 (Experimental)
  Interventions: Drug: Cetrorelix 78+78
- Cetrorelix 78 + Placebo (Experimental)
  Interventions: Drug: Cetrorelix 78 + Placebo
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cetrorelix 78+78 — Cetrorelix 78 mg combining Week 0 (52 mg) and Week 2 (26 mg) + 78 mg combining Week 26 (52 mg) and Week 28 (26 mg)
  Arms: Cetrorelix 78+78
Drug: Cetrorelix 78 + Placebo — Cetrorelix 78 mg combining Week 0 (52 mg) and Week 2 (26 mg) + Placebo on Week 26 and Week 28
  Arms: Cetrorelix 78 + Placebo
Other: Placebo — Placebo on Week 0, Week 2, Week 26 and Week 28
  Arms: Placebo

SUMMARY:
Benign Prostatic Hypertrophy (BPH) is a common and bothersome condition of aging men. It is characterized by an enlargement of the prostate occurring in human male over the age of 50 which increases in prevalence with age, and among those aged 50 to 80, about 40% report moderate or severe urinary symptoms of prostatism. The aim of treatment is to improve patients' quality of life which primarily depends on the severity of the symptoms of BPH. Current treatments of BPH have a benefit / risk ratio which leaves room for improvement.

For this study, study medication (Cetrorelix pamoate or placebo) is administered by injection in the buttocks (Intramuscular). All patients completing the double-blind portion (Week 0 to 52) are eligible to receive the active drug during the open-label part of the study (Week 52 to 90).

ELIGIBILITY:
Inclusion Criteria:

* Benign Prostatic Hyperplasia, based on medical history
* Voiding symptoms

Exclusion Criteria:

* Urgent need for prostate surgery or prior surgical treatment of the prostate or bladder
* Major organ dysfunction
* Eczema (atopic dermatitis) treated during the last 6 months
* Current or recent treatment with sexual hormone drugs or 5 α reductase inhibitors or botulinum toxin type a (Botox) within the last 6 months prior randomization or with α blockers or saw palmetto within the last 6 weeks prior to randomization
* Urologic disorders including neurogenic bladder dysfunction due to diabetes mellitus or documented neurologic disorder, urethral stricture disease or history of pelvic radiation therapy
* History of acute obstructive, infectious, or neurological disorders of the genitourinary tract within the last 3 months

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans MJ Debruyne, M.D., Study Chair — Andros Mannenkliniek, Arnhem, The Netherlands
Locations (54):
- Belarus (3):
  - 19th Central Regional Policlinic, Urology department, Minsk
  - 4th City Hospital, Minsk
  - Minsk Regional Clinical Hospital, Clinic of Urology, Minsk
- Bulgaria (5):
  - University multiprofil Hospital of Active Treatment "Sveti Georgi", Urology Department, Plovdiv
  - Aleksandrovska Hospital, Kidney Transplantation Department, Sofia
  - Aleksandrovska Hospital, Oncourology Department, Sofia
  - National Central Hospital for Active Treatment of Oncology JSC, Sofia
  - Multiprofil Hospital "Sveta Anna", Urology Department, Varna
- Czechia (9):
  - Privat urological ambulance, Besenov
  - Health Center SANUS, Hradec Králové
  - Privat urological ambulance, Pilsen
  - Urocentrum Prague, Out-Patient Clinic of Urology, Prague
  - 1st Medical Faculty of Charles University, Deputy Department and Clinic of Urology, Prague
  - Urological center Uro-Santé Brumlovka, Prague
  - Androgeos Clinic, Prague
  - Policlinic Pod Marjánkou 12, Urological Department, Prague
  - Faculty hospital Na Bulovce, Prague
- France (5):
  - Hopital Henri Mondor Service Urologie, Créteil
  - CHU Hôpital Claude Huriez, Lille
  - Hopital Edouard Heriot Service Urologie, Lyon
  - Hopital René Dubos Service Urologie 6, Pontoise
  - C.H.U Rangueil, Service d'Urologie, Toulouse
- Germany (9):
  - Pan-Klinik Urologie, Cologne
  - Urologische Gemeinschaftspraxis Rulf/Langhorst, Erkrath
  - Urologische Praxisgemeinschaft Frankfurt Höchst, Frankfurt
  - Urologische Praxis, Marburg
  - Urologische Praxis, Münster
  - Urologische Klinik, Ev. Krankenhaus Oberhausen, Oberhausen
  - Klinikum Offenbach GmbH, Klinik für Urologie, Offenbach
  - Asklepios Klinik Seligenstadt, Seligenstadt
  - Praxis Filipas, Wiesbaden
- Italy (5):
  - University of Bari, Department of Urology, Bari
  - Irccs Ospedale San Raffaele Milano, Università Vita Salute-San Raffaele, Milan
  - Università Federico II Napoli, Naples
  - Università Federico II Napoli, Napoli
  - University of Padova, Department of Urology, Padua
- Netherlands (8):
  - Gelre Ziekenhuizen, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Andros Mannenkliniek, Arnhem
  - Atrium Medisch Centrum, Heerlen
  - Andros Mannenkliniek, Leiden
  - Andros Mannenkliniek, Maastricht
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Streekziekenhuis Koningin Beatrix, Winterswijk
- Urology Clinic Skopje, Skopje, North Macedonia
- Romania (5):
  - S.C. Uro Andro Med Srl, Bucharest
  - Spitalul Clinic de Urgenta "Sf. Ioan", Clinica Urologie, Bucharest
  - Spitalul Clinic de Urologie "Prof. Dr. Th. Burghele", Bucharest
  - Clinica Chirurgie Urologica si Transplant Renal, Bucharest
  - Centrul Medical "Sf. Pantelimon", Pantelimon
- United Kingdom (4):
  - Leighton Hospital, Clinical Trials Dept., Michael Heal Unit, Crewe, Cheshire
  - Bristol Royal Infirmary, Urology Research Unit, Bristol
  - Leicester General Hospital, Urology Section, Leicester
  - Freeman Hospital, Urology Clinic, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetrorelix 78+78: 78 mg combining Week 0 (52 mg) and Week 2 (26 mg) + 78 mg combining Week 26 (52 mg) and Week 28 (26 mg)
- CET 78+Placebo: 78 mg combining Week 0 (52 mg) and Week 2 (26 mg) + Placebo on Week 26 and Week 28.
- Placebo: Placebo on Week 0, 2, 26 and 28.
Period: Overall Study
Arm/Group | Cetrorelix 78+78 | CET 78+Placebo | Placebo
Started | 212 | 106 | 102
Completed | 178 | 96 | 82
Not Completed | 34 | 10 | 20
Not completed — Adverse Event | 9 | 1 | 6
Not completed — Lack of Efficacy | 5 | 1 | 3
Not completed — Withdrawal by Subject | 7 | 3 | 3
Not completed — Protocol Violation | 5 | 3 | 4
Not completed — Other | 8 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetrorelix 78+78 | CET 78+Placebo | Placebo | Total
Number analyzed (Participants) | 212 | 106 | 102 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 101 | 45 | 37 | 183
  >=65 years | 111 | 61 | 65 | 237
Age Continuous [Mean (Standard Deviation); unit: years] | 66.58 (8.16) | 66.50 (7.29) | 67.72 (7.17) | 66.83 (7.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 212 | 106 | 102 | 420
Region of Enrollment [Number; unit: participants]
  France | 0 | 1 | 0 | 1
  Belarus | 37 | 18 | 18 | 73
  Czech Republic | 33 | 15 | 19 | 67
  Macedonia, The Former Yugoslav Republic of | 6 | 3 | 3 | 12
  Romania | 54 | 28 | 26 | 108
  Bulgaria | 41 | 20 | 20 | 81
  Germany | 15 | 7 | 6 | 28
  Netherlands | 23 | 13 | 10 | 46
  United Kingdom | 1 | 0 | 0 | 1
  Italy | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS)
Description: IPSS score of BPH symptoms based on a patient questionnaire assessing 7 items (incomplete voiding, frequency, intermittency, urgency, weak stream, hesitancy, nocturia) on a scale from 0 (best) to 5 (worst); total overall score range: 0 points (best) to 35 points (worst)
Time Frame: Baseline and 52 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cetrorelix 78+78 | CET 78+Placebo | Placebo
Number analyzed (Participants) | 207 | 104 | 100
Units on a scale | -6.2 (5.68) | -5.1 (5.18) | -5.7 (6.04)
Statistical Analysis 1: Comparison: Cetrorelix 78+78 vs Placebo; Test type: Superiority or Other; p = 0.371, ANOVA; Mean Difference (Final Values) = -0.592, 95% CI 2-sided [-1.894 to 0.709], Standard Error of Mean 0.662
Statistical Analysis 2: Comparison: CET 78+Placebo vs Placebo; Test type: Superiority or Other; p = 0.3253, ANCOVA; Mean Difference (Final Values) = 0.711, 95% CI 2-sided [-0709 to 2.132], Standard Error of Mean 0.722
Statistical Analysis 3: Comparison: Cetrorelix 78+78 vs CET 78+Placebo; Test type: Superiority or Other; p = 0.0333, ANCOVA; Mean Difference (Final Values) = -1.324, 95% CI 2-sided [-2.542 to -0.106], Standard Error of Mean 0.620

ADVERSE EVENTS:
Arm/Group | Cetrorelix 78+78 | CET 78+Placebo | Placebo
Serious Adverse Events (participants affected / at risk) | 8/212 | 7/106 | 5/102
Other Adverse Events (participants affected / at risk) | 10/212 | 5/106 | 6/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetrorelix 78+78 (N=212) | CET 78+Placebo (N=106) | Placebo (N=102)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster ophtalmic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infarction (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infartion (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetrorelix 78+78 (N=212) | CET 78+Placebo (N=106) | Placebo (N=102)
Influenza (Infections and infestations) | 10 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days